CLINICAL TRIAL: NCT04124315
Title: Using Smartphone Sensor Technology to Characterize Ambulatory Patterns of Participants With Peripheral Artery Disease
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: SON-2019-28208
Record Dates: First submitted 2019-10-10; First posted 2019-10-11 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral artery disease; accelerometer; smartphone; supervised exercise therapy
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Accelerometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PAD Patients Completing SET: This single-group study includes patients with peripheral artery disease (PAD) who are completing a physician-prescribed supervised exercise training (SET) program.
  Interventions: Other: Accelerometry; Other: Daynamica app

INTERVENTIONS:
Other: Accelerometry — Patients will be given accelerometers at this visit and informed on how to use them (e.g., wear on the ankle during waking hours, upright, etc).
Other: Daynamica app — Participants will be asked to record location/activity on the app in order to characterize activity patterns both inside and outside of the hospital SET setting.

SUMMARY:
The investigators plan to use smartphone and wearable sensor technology to characterize the activity patterns of participants with peripheral artery disease (PAD) (n=24) participating in a 12-week supervised exercise training (SET) program, and incorporate the resulting data into a web-based dashboard for participants and study staff.

DETAILED DESCRIPTION:
Participants in the proposed study will be current clinical participants in the SET program within Fairview. Participants will have a diagnosis of PAD and be ≥40 years of age (participants are diagnosed before they are referred to the SET program). Rate limiting comorbidities not associated with vascular disease (e.g., severe chronic obstructive pulmonary disease) will be exclusionary (for example). Age, sex, race, ethnicity, educational status, and smoking status at baseline will be recorded from cardiac rehabilitation intake forms. Eligible participants will be identified by study staff reviewing electronic medical records of patients who are enrolling into the SET program. University of Minnesota staff will travel to the urban and rural clinical rehabilitation sites to obtain informed consent at the participants first SET visit. They will then provide participants instructions and training for how to use the smartphone and app.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of atherosclerotic PAD and referred to hospital-based SET
* Ability to complete an evaluation of physical function and walk on a treadmill
* Resting ankle-brachial index (ABI) of ≤0.90 or stenosis ≥50% in a peripheral vessel or those with lifestyle limiting vascular-related claudication
* Those with a resting ABI of 0.91-0.99 (borderline) who have completed an exercise-ABI assessment with a >20% drop compared to resting values
* Those with ABI >1.40 who have had an abnormal toe-brachial index of ≤0.70

Exclusion Criteria:

* Lower extremity amputation(s) which interfere(s) with walking on the treadmill.
* Individuals with critical limb ischemia defined by ischemic rest pain or ischemic ulcers/gangrene on the lower extremities
* PAD of non-atherosclerotic nature (e.g., fibromuscular dysplasia, irradiation, endofibrosis)
* Females who are pregnant
* Coronary artery bypass grafts or major surgical procedures within 6 months prior to screening
* Individuals whose walking exercise is primarily limited by symptoms of chronic obstructive pulmonary disease, angina, or heart failure
* Individuals who have had a myocardial infarction within 3 months prior to screening
* Individuals who have had a transient ischemic attack or stroke 3 months prior to screening
* Individuals with uncontrolled hypertension (≥180 systolic or ≥100 diastolic resting blood pressure) during screening
* Poorly controlled diabetes defined as glycated hemoglobin >12%
* Abnormal results of blood work not conducive to safely participating in an exercise trial (e.g., anemic, electrolyte abnormalities)
* Inability to speak English
* Other clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurological, psychiatric, immunological, gastrointestinal, hematological, or metabolic disease that is, in the opinion of the study team, not stabilized or may otherwise confound the results of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PAD patients completing exercise training in the cardiac rehab programs in the Fairview Health System. The five Fairview hospital-based sites are located at urban and rural sites within and outside of the Twin Cities metropolitan area: Riverside (Minneapolis/St. Paul, MN), Southdale (Edina, MN), Ridges (Burnsville, MN), Lakes (Wyoming, MN), and Northland (Princeton, MN).
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in The Walking Impairment Questionnaire (WIQ) Distance Subcategory | 12 weeks
  In the Walking Impairment Questionnaire distance subcategory, participants are asked to rate the degree of difficulty walking specific distances on a scale from 0 to 4. A score of 0 indicates the inability to walk the distance specified by the question while a score of 4 represents no difficulty. The graded sub-score is multiplied by a pre-specified weight for each sub-category: distance, speed, and number of flights of stairs. The products of these subscores are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (inability to perform item) to 100 (no difficulty in performing item).
Change in The Walking Impairment Questionnaire (WIQ) Speed Subcategory | 12 weeks
  In the Walking Impairment Questionnaire speed subcategory, participants are asked to rate the degree of difficulty walking one block at specific speeds, ranging from walking slowly to jogging, on a scale from 0 to 4. A score of 0 indicates the inability to walk the distance specified by the question while a score of 4 represents no difficulty. The graded sub-score is multiplied by a pre-specified weight for each sub-category: distance, speed, and number of flights of stairs. The products of these subscores are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (inability to perform item) to 100 (no difficulty in performing item).
Change in The Walking Impairment Questionnaire (WIQ) Stair-Climbing Subcategory | 12 weeks
  In the Walking Impairment Questionnaire stair-climbing subcategory, participants are asked to rate the degree of difficulty climbing a specified number of stair flights, ranging from 1 to 3 stair flights, on a graded scale of 0 to 4. A score of 0 indicates the inability to climb the flights specified by the question while a score of 4 represents no difficulty. The graded sub-score is multiplied by a pre-specified weight for each sub-category: distance, speed, and number of flights of stairs. The products of these subscores are summed and divided by the maximum possible score to obtain a percent score, ranging from 0 (inability to perform item) to 100 (no difficulty in performing item).
Change in SF-36 Physical Component Summary | 12 weeks
  The SF-36 has eight scaled subscores (Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health). These subscores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability.
Change in SF-36 Mental Component Summary | 12 weeks
  The SF-36 has eight scaled subscores (Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, Mental health). These subscores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability.
Peripheral Artery Disease Quality of Life (PADQOL) questionnaire | 12 weeks
  PADQOL is a 38-item survey assessing the quality of life of PAD patients. Items are scored on a scale of 1 (strongly agree) to 6 (strongly disagree). Total scores are sums of all 38 items with a range of 38 (normal quality of life) to 228 (quality of life is severely impaired).

SECONDARY OUTCOMES:
Change in Ankle-Brachial Index (ABI) Assessment | 12 weeks
  The Ankle Brachial Index (ABI) calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressure at the arm. Values between 1.0 and 1.4 are considered clinically normal while lower scores indicate greater progression of vascular disease with scores less than 0.5 indicating severe PAD.
Change in Six-Minute Walk Test (6-MWT) Maximal Distance | 12 weeks
  Participants will walk in a 50-foot corridor at the hospital. Maximal walking distance achieved in 6 minutes is recorded in feet. Decreased walking distance indicates increased impairment due to PAD.
Change in Six-Minute Walk Test (6-MWT) Claudication Onset Time | 12 weeks
  Participants will walk in a 50-foot corridor at the hospital. Claudication onset time is recorded in seconds. Decreased time for claudication onset indicates increased impairment due to PAD.
Change in Six-Minute Walk Test (6-MWT) Claudication Onset Distance | 12 weeks
  Participants will walk in a 50-foot corridor at the hospital. Claudication onset distance is recorded in feet. Decreased walking distance before claudication onset indicates increased impairment due to PAD.
Short Physical Performance Battery (SPPB) | 12 weeks
  The SPPB is a group of measures including balance, gait speed, and chair stand. In the balance sub test, patients are awarded points for holding a position for a longer period of time. The balance sub score is a summed value ranging from 0 to 4.
  In the gait speed sub test, patients are awarded points for walking a set distance in less time. The gait speed sub score ranges from 1 (time > 8.7 sec) to 4 (time < 4.82 sec) for a 4-meter distance and 1 (time > 6.52 sec) to 4 (time < 3.62 sec) for the 3-meter distance.
  In the chair stand sub test, patients are asked to stand from a sitting position. The chair stand sub score ranges from 0 (unable to complete 5 chair stands or completes stand in >60 sec) to 4 (chair stand time is 11.19 sec of less).
  The SPPB total score is an unweighted sum of the 3 sub scores, with possible total scores ranging from 1 to 12. Higher scores indicate better function.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Mays, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No